CLINICAL TRIAL: NCT00472719
Title: A Phase 1B Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Adenoviral Serotype 35 (rAd35) and Serotype 5 (rAd5) HIV-1 Vaccines When Given in Heterologous Prime-Boost Regimens or as a Boost to a Recombinant DNA Vaccine in Healthy, HIV-1-Uninfected Adult Participants With Pre-Existing Immunity to Adenovirus Serotype 5 Infection
Brief Title: Safety of and Immune Response to a DNA HIV Vaccine Followed By Boosting With One of Two Serotypes of Adenoviral Vector HIV Vaccine in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: HIV Vaccine Trials Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HVTN 072; 10517 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: HIV Seronegativity; HIV Preventive Vaccine; Adenovirus
MeSH Terms: conditions — HIV Infections; Adenoviridae Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants in this group will receive an injection of the adenoviral vector vaccine VRC-HIVADV027-00VP at study entry and an injection of VRC-HIVADV038-00-VP at Month 3. There will be 9 study visits for this arm.
  Interventions: Biological: VRC-HIVADV027-00-VP; Biological: VRC-HIVADV038-00-VP
- 2 (Experimental): Participants in this group will receive an injection of VRC-HIVADV038-00-VP at study entry and an injection of VRC-HIVADV027-00-VP at Month 3. There will be 9 study visits for this group.
  Interventions: Biological: VRC-HIVADV027-00-VP; Biological: VRC-HIVADV038-00-VP
- 3 (Experimental): Participants in this group will receive an injection of the VRC-HIVDNA044-00-VP vaccine at study entry and Months 1 and 2, followed by an injection of VRC-HIVADV027-00-VPat Month 6. There will be 13 study visits for this group.
  Interventions: Biological: VRC-HIVADV027-00-VP; Biological: VRC-HIVDNA044-00-VP
- 4 (Experimental): Participants in this group will receive an injection of VRC-HIVDNA044-00-VP at study entry and Months 1 and 2, followed by an injection of VRC-HIVADV038-00-VP at Month 6. There will be 13 study visits for this group.
  Interventions: Biological: VRC-HIVADV038-00-VP; Biological: VRC-HIVDNA044-00-VP

INTERVENTIONS:
Biological: VRC-HIVADV027-00-VP — Adenoviral vector booster vaccine
  Arms: 1; 2; 3
Biological: VRC-HIVADV038-00-VP — Adenovirus vector booster vaccine
  Arms: 1; 2; 4
Biological: VRC-HIVDNA044-00-VP — Experimental, multiclade, multigene HIV DNA vaccine
  Arms: 3; 4

SUMMARY:
The purpose of this study is to determine the safety of and immune response to an experimental DNA HIV vaccine followed by boosting with either an experimental adenoviral vector HIV vaccine of serotype 5 or 35 in HIV uninfected adults. This study will also determine the safety of and immune response to an adenoviral vector HIV vaccine of serotype 5 followed by a booster of an adenoviral vector of serotype 35, or vice versa, in HIV uninfected adults.

DETAILED DESCRIPTION:
The worldwide HIV/AIDS epidemic may only be controlled through development and utilization of a safe and effective vaccine that will prevent HIV infection. Vaccines using a DNA plasmid to prime the response to an adenoviral vector boost are currently being developed. Due to high prevalence of pre-existing immunity to adenovirus serotype Ad5 in the developing world, this study will evaluate boosting with a different serotype, Ad35, as compared to boosting with the Ad5 serotype. This study will also test the effect of the order of administration of recombinant adenoviral vector HIV vaccines when administered without the DNA plasmid vaccine. Two arms of this study will evaluate the safety and immunogenicity of the experimental multiclade, multigene HIV DNA vaccine VRC-HIVDNA044-00-VP, followed by a similarly structured adenovirus vector vaccine boost (either VRC-HIVADV027-00-VP or VRC-HIVADV038-00-VP), in HIV uninfected adults. To determine the effect of pre-existing Ad5 or Ad35 immunity, the other two arms will test the safety and immunogenicity of receiving either VRC-HIVADV027-00-VP followed by VRC-HIVADV038-00-VP, or vice versa.

Each volunteer will participate in the study for at least 6 months. Participants will be randomly assigned to one of four groups and will receive either an experimental vaccine or placebo at each vaccination visit. Group 1 participants will receive an injection of the adenoviral vector vaccine VRC-HIVADV027-00-VP at study entry and an injection of VRC-HIVADV038-00-VP at Month 3. Group 2 participants will receive an injection of the adenoviral vector vaccine VRC-HIVADV038-00-VP at study entry and an injection of VRC-HIVADV027-00-VP at Month 3. Group 3 participants will receive an injection of the VRC-HIVDNA044-00-VP vaccine at study entry and Months 1 and 2, followed by an injection of VRC-HIVADV027-00-VP at Month 6. Group 4 participants will receive an injection of the DNA HIV vaccine at study entry and Months 1 and 2, followed by an injection of VRC-HIVADV038-00-VP at Month 6.

For Groups 1 and 2, there will be 9 study visits. For Groups 3 and 4, there will be 13 study visits. Medication history, assessment of intercurrent illness and adverse effects, and HIV and pregnancy prevention counseling will occur at all visits. A medical history, a physical exam, HIV testing and counseling and blood and urine collection will occur at selected visits. Participants will also be asked to complete social impact and HIV testing and history questionnaires at selected visits.

As of 11/19/07 enrollment and vaccinations have been discontinued. Participants who have already been enrolled have been told which vaccinations they received and will be followed for a total of 5 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 and -2 uninfected
* Have access to a participating HIV Vaccine Trials Unit (HVTU) and willing to be followed for the duration of the study
* Willing to receive HIV test results
* Good general health
* Pre-existing adenovirus 5 (Ad5) neutralizing antibody titer of 1:1000 ratio or greater
* Willing to use acceptable forms of contraception from at least 21 days prior to enrollment through the duration of the study

Exclusion Criteria:

* HIV vaccines in prior HIV vaccine trial
* Immunosuppressive medications within 168 days prior to first study vaccine administration
* Blood products within 120 days prior to first study vaccine administration
* Immunoglobulin within 60 days prior to first study vaccine administration
* Live attenuated vaccines within 30 days prior to first study vaccine administration
* Investigational research agents within 30 days prior to first study vaccine administration
* Subunit or killed vaccines within 14 days prior to first study vaccine administration
* Current anti-tuberculosis prophylaxis or therapy
* Clinically significant medical condition, abnormal physical exam findings, abnormal laboratory results, or past medical history that may affect current health. More information about this criterion can be found in the protocol.
* Any medical, psychiatric, or social condition that would interfere with the study.
* Serious adverse reaction to vaccines. Participants who have had an adverse reaction to pertussis vaccine as a child are not excluded.
* Autoimmune disease or immunodeficiency
* Active syphilis infection. Participants with fully treated syphilis at least 6 months prior to study entry are not excluded.
* Unstable asthma. More information about this criterion can be found in the protocol.
* Diabetes mellitus type 1 or 2. Participants with a history of isolated gestational diabetes are not excluded.
* Absence of thyroid or thyroid disease requiring treatment
* Serious angioedema within the past 3 years or requiring medication within 2 years of study entry
* Body mass index (BMI) of 40 or less OR BMI of 35 or less if certain other criteria apply. More information about these criteria can be found in the protocol.
* Uncontrolled hypertension
* Bleeding disorder
* Cancer. Participants with surgically removed cancer that is unlikely to recur are not excluded.
* Seizure disorder
* Absence of spleen
* Certain abnormal laboratory values
* Mental illness that would interfere with compliance with the protocol
* Other conditions that, in the judgment of the investigator, would interfere with the study
* Pregnant or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2007-08; Primary Completion 2008-07 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of HIV-1 recombinant Clade A env DNA, rAd5, and rAd35 vaccines in participants with pre-existing immunity to Ad5 | at 9 to 12 months
Magnitude and frequency of immune responses between the adenoviral vaccines following DNA prime, assessed by enzyme-linked immunospot (ELISpot) responses, intracellular cytokine staining (ICS) T-cell responses, and HIV-1 antibody assays | at 4 weeks following fourth vaccination
Immunogenicity of recombinant HIV-1 Clade A env rAd35 vaccine following a recombinant rAd5 prime, assessed by ELISpot responses, ICS T-cell responses, and HIV-1 antibody assays | at 4 weeks following the second vaccination
Immunogenicity of recombinant HIV-1 Clade A env rAd5 vaccine following a recombinant rAd35, assessed by ELISpot responses, ICS T-cell responses, and HIV-1 antibody assays | at 4 weeks following the second vaccination

SECONDARY OUTCOMES:
Rank of HIV-1 rAd5/rAd35, rAd35/rAd5, DNA/rAd5, and DNA/rAd35 regimens based on ELISpot responses, ICS T-cell responses, and HIV-1 antibody assays | at 4 weeks after second vaccination for Groups 1 and 2, and at 4 weeks after fourth vaccination for Groups 3 and 4
Immunogenicity of HIV-1 rAd35 vaccine given as a prime assessed by ELISpot responses, ICS T-cell responses, and HIV-1 antibody assays | at 4 weeks following first vaccination
Immunogenicity of HIV-1 rAd5 vaccine given as a prime, assessed by ELISpot responses, ICS T-cell responses, and HIV-1 antibody assays | at 4 weeks following first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Fuchs, MD, MPH, Study Chair — San Francisco Department of Public Health, University of California, San Francisco
Locations (7):
- United States (7):
  - Alabama Vaccine CRS, Birmingham, Alabama
  - Bridge HIV CRS, San Francisco, California
  - Columbia P&S CRS, New York, New York
  - New York Blood Center CRS, New York, New York
  - University of Rochester Vaccines to Prevent HIV Infection CRS, Rochester, New York
  - Vanderbilt Vaccine (VV) CRS, Nashville, Tennessee
  - Seattle Vaccine and Prevention CRS, Seattle, Washington

REFERENCES:
- [Background] Barouch DH, Nabel GJ. Adenovirus vector-based vaccines for human immunodeficiency virus type 1. Hum Gene Ther. 2005 Feb;16(2):149-56. doi: 10.1089/hum.2005.16.149. PMID 15761255
- [Background] Barouch DH, Pau MG, Custers JH, Koudstaal W, Kostense S, Havenga MJ, Truitt DM, Sumida SM, Kishko MG, Arthur JC, Korioth-Schmitz B, Newberg MH, Gorgone DA, Lifton MA, Panicali DL, Nabel GJ, Letvin NL, Goudsmit J. Immunogenicity of recombinant adenovirus serotype 35 vaccine in the presence of pre-existing anti-Ad5 immunity. J Immunol. 2004 May 15;172(10):6290-7. doi: 10.4049/jimmunol.172.10.6290. PMID 15128818
- [Background] Cohen P. Immunity's yin and yang. A successful vaccine must first avoid being eliminated by pre-existing immunity before it can promote a protective immune response. IAVI Rep. 2006 Jan-Feb;10(1):1-5. No abstract available. PMID 16625717
- [Background] Lemckert AA, Sumida SM, Holterman L, Vogels R, Truitt DM, Lynch DM, Nanda A, Ewald BA, Gorgone DA, Lifton MA, Goudsmit J, Havenga MJ, Barouch DH. Immunogenicity of heterologous prime-boost regimens involving recombinant adenovirus serotype 11 (Ad11) and Ad35 vaccine vectors in the presence of anti-ad5 immunity. J Virol. 2005 Aug;79(15):9694-701. doi: 10.1128/JVI.79.15.9694-9701.2005. PMID 16014931
- [Background] Wu L, Kong WP, Nabel GJ. Enhanced breadth of CD4 T-cell immunity by DNA prime and adenovirus boost immunization to human immunodeficiency virus Env and Gag immunogens. J Virol. 2005 Jul;79(13):8024-31. doi: 10.1128/JVI.79.13.8024-8031.2005. PMID 15956548